CLINICAL TRIAL: NCT03522220
Title: Augmentation of Neuronal Network Plasticity in Schizophrenia
Acronym: SCZ
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Basic Science
Other Study IDs: SFB936 C7
Record Dates: First submitted 2018-04-30; First posted 2018-05-11 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Schizophrenia; Healthy
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 3D Super Mario Game Condition (Experimental): 3D navigation video game intervention
  Interventions: Behavioral: 3D navigation video game intervention
- 2D Super Mario Game Condition (Active Comparator): Video game intervention without 3D navigation
  Interventions: Behavioral: video game intervention without 3D navigation
- Kindle Device (Active Comparator): No 3D navigation
  Interventions: Behavioral: No 3D navigation

INTERVENTIONS:
Behavioral: 3D navigation video game intervention — Participants intensively train with a video game (Super Mario DS)
  Arms: 3D Super Mario Game Condition
Behavioral: video game intervention without 3D navigation — Participants train with a video game (Super Mario Bros)
  Arms: 2D Super Mario Game Condition
Behavioral: No 3D navigation — Participants read on a kindle device (control group)
  Arms: Kindle Device

SUMMARY:
Current pathophysiological models of schizophrenia focus on disconnectivity of distributed neuronal systems to explain the multitude of psychic symptoms. However, therapeutic strategies targeting this specific pathobiology are lacking. Our recent work provides strong evidence that complex video-game training interventions facilitate fronto-hippocampal structural and functional connectivity within 2 months in healthy subjects. The planned project transfers this knowledge into a training study in schizophrenic patients to counteract disease-related disconnectivity. Underlying mechanisms and behavioral effects are extensively parametrized by resting state functional magnetic resonance imaging (fMRI), diffusion tensor imaging (DTI), spectroscopy and clinical short- and long-term outcome.

ELIGIBILITY:
Inclusion Criteria:

* clinically stabilized
* at least one schizophrenic episode in their lives
* International Classification of Diseases 10 (ICD-10) F20.x (and F25)

Exclusion Criteria:

* clinically relevant anemia
* MRI contraindication
* earlier electroconvulsive shock treatment
* significant somatic or neurological disease
* significant alcohol or substance abuse in the year before
* more than 1h video games per day more than 6 months before study start
* simultaneous major psychiatric disease (if symptomatic in the foreground)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-09-01 (Actual); Primary Completion 2019-07-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
T1 - MRI | 2 months (= training time and 2 months after training end)
  The investigators look for structural volume changes in T1 images (MRI) specifically in the hippocampus and prefrontal areas due to training
Cognition - Spatial Orientation | 2 months (= training time and 2 months after training end)
  The investigators look for changes in cognition specifically regarding spatial orientation (MATRICS, computer tests measuring spatial orientation with and without external cue) due to training.
Positive & Negative Symptoms in patients | 2 months (= training time and 2 months after training end)
  The investigators look for changes in positive and negative symptoms (PANSS) due to training.

SECONDARY OUTCOMES:
Resting State fMRI | 2 months (= training time and 2 months after training end)
  The investigators look for blood oxygen level dependency (BOLD) changes in resting state fMRI specifically in the Hippocampus and Prefrontal Areas due to the training
Spectroscopy - glutamate | 2 month (= training time and 2 month after training end)
  The investigators look for glutamate concentration changes in the hippocampus due to the training
Diffusion Tensor Imaging (DTI) | 2 month (= training time and 2 month after training end)
  The investigators look for structural connectivity changes in DTI images due to the training
Biomarkers (BDNF & interleukin 1 & 6) | 2 month (= training time and 2 month after training end)
  The investigators look for plasticity induced changes in biomarkers (interleukin1 and 6 and BDNF [brain-derived neurotrophic factor]) due to training

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinic Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://www.sfb936.net/thematic-area-c